CLINICAL TRIAL: NCT00497562
Title: Exploratory Study to Investigate the Efficacy and Safety of Recombinant Growth Hormone as Add-on Treatment in Patients With Severe Fibromialgia
Brief Title: Growth Hormone as Add-on Treatment in Severe Fibromyalgia With Low IGF-1 Serum Levels (56 Characters)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Medico Teknon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FibTek-0301; 03-0453 (AGEMED)
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Fibromyalgia; Growth Hormone Deficiency
Keywords: Fibromyalgia; growth hormone; IGF-1; FIQ
MeSH Terms: conditions — Fibromyalgia; Dwarfism, Pituitary | interventions — Amitriptyline; Fluoxetine; Tramadol; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: sc recombinant growth hormone + amitriptyline, fluoxetine and tramadol (treated group)
Drug: amitriptyline, fluoxetine and tramadol alone (control group)

SUMMARY:
There are evidences of functional growth hormone (GH) deficiency, expressed by means of low serum levels of insulin-like growth factor 1 (IGF-1), in a subset of fibromyalgia patients. The efficacy of low GH doses versus placebo has been demonstrated in this population. We assessed the efficacy and safety of GH added to standard therapy compared to standard therapy alone in the treatment of severe, prolonged and well-treated fibromialgya patients with low IGF-1 levels.

ELIGIBILITY:
Inclusion Criteria:

* Women greater than 18 years old with severe fibromyalgia and abnormally low IGF-1 levels included in a rehabilitation and psychological program and stable under standard intensive treatment for at least 6 months.
* All patients fulfilled the 1990 ACR diagnostic criteria (1) and had an IGF-1 level <250 ng/mL (or 1 standard deviation bellow the mean value corresponding to age and body surface according to laboratory reference value).
* Other inclusion criteria were duration of fibromyalgia of 1 year or greater, pain in at least 16 (8 bilateral) of the 18 tender points and a score in the FIQ > 75.
* The study was conducted in accordance with the Declaration of Helsinki and received the local institutional review board and Spanish Drug Agency (nº03-0456) approvals. All patients gave written informed consent prior to their inclusion in the study.

Exclusion Criteria:

* Disabling physical or mental status
* Previous or current malignancies, either active or inactive
* Intracranial space occupying lesion
* Any relevant endocrine disorder including diabetes mellitus
* History of another pituitary disorder
* Previous treatment with growth hormone
* Other systemic or joint inflammatory rheumatic conditions; and
* Known to be hypersensitive to somatropin or any of the excipients.
* Pregnant women, nursing mothers, or women with childbearing potential not using adequate contraceptive methods were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-05; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
reduction number of tender points (paired) | one year treatment

SECONDARY OUTCOMES:
improvement in FIQ, EQ-5D , analogic visual scales (1). Safety (2). | one year

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Cuatrecasas, MD, Principal Investigator — CM Teknon Endocrinology Head Department; Albert Nadal, MD, Study Chair — CM Teknon Rheumatology Head Department
Locations (1):
- Endocrinology Department CM Teknon, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Bennett RM, Clark SC, Walczyk J. A randomized, double-blind, placebo-controlled study of growth hormone in the treatment of fibromyalgia. Am J Med. 1998 Mar;104(3):227-31. doi: 10.1016/s0002-9343(97)00351-3. PMID 9552084
- [Background] Leal-Cerro A, Povedano J, Astorga R, Gonzalez M, Silva H, Garcia-Pesquera F, Casanueva FF, Dieguez C. The growth hormone (GH)-releasing hormone-GH-insulin-like growth factor-1 axis in patients with fibromyalgia syndrome. J Clin Endocrinol Metab. 1999 Sep;84(9):3378-81. doi: 10.1210/jcem.84.9.5982. PMID 10487713
- [Derived] Cuatrecasas G, Riudavets C, Guell MA, Nadal A. Growth hormone as concomitant treatment in severe fibromyalgia associated with low IGF-1 serum levels. A pilot study. BMC Musculoskelet Disord. 2007 Nov 30;8:119. doi: 10.1186/1471-2474-8-119. PMID 18053120